CLINICAL TRIAL: NCT05090007
Title: Imaging of Injury Mechanism and Interaction of Intestinal Bacteria in Children With Mild Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xi'an Jiaotong University (Other); The Second Affiliated Hospital and Yuying Childern's Hospital of Wenzhou Medical University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 82071993
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: MTBI - Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury, MRI, gut microbiota
MeSH Terms: conditions — Brain Concussion | interventions — Magnetic Resonance Imaging; Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gut microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mTBI: A TBI is caused by a bump, blow, or jolt to the head that disrupts the normal function of the brain. Not all blows or jolts to the head result in a TBI.
  Interventions: Device: magnetic resonance image; Other: gut microbiota
- HC: Healthy controls
  Interventions: Device: magnetic resonance image; Other: gut microbiota

INTERVENTIONS:
Device: magnetic resonance image — Imaging data were collected in a strong magnetic field
Other: gut microbiota — gut microbiota

SUMMARY:
Traumatic brain injury (TBI) is the leading cause of disability in children and young adults. Children with moderate to severe TBI are typically at risk of poor functional outcome in terms of neurocognitive impairment and behavior problems. Neurocognitive impairments include deficits in attention and working memory, learning and memory, and executive functioning, whereas behavior problems include anxiety, depression and aggression. Neuroimaging techniques based on multi-modal magnetic resonance image (MRI) can detect the structural and functional brain abnormalities objectively and sensitively. Recent evidence indicates that even after mild TBI, children with risk factors for intracranial pathology are at risk of poor neurocognitive and behavioral outcome.Meanwhile, recently, the concept of "gut-brain axis" has been proposed and hint gut microbiota could shape the brain. Some studies have emphasized that human gut microbiota plays an important role in the pathogenesis and development of TBI. However, how the gut affects the brain in patients with TBI is unclear. Thus, combining analysis of neuroimaging and "gut-brain axis" will provide more information for finding the risk factors and imaging diagnostic markers of brain impairment in TBI. It will also helpful for explaining the underlying mechanisms of brain impairment in TBI, providing an objective basis for clinical diagnosis and prediction of the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* age 6-14 years at time of recruitment.
* hospital admission with a clinical diagnosis of TBI for inclusion in the TBI group
* GCS = 15-13.
* loss of consciousness duration≤30 min.
* post-traumatic amnesia duration ≤1 h.

Exclusion Criteria:

* previous TBI.
* visual or auditory disorder interfering with neurocognitive testing.
* current neurological condition affecting the central nervous system with known effects on neurocognitive functioning, other than TBI.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All of the patients of mTBI group are in-patients and out-patients in the nephrology department from three research centers. The subjects of control group are recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline brain structure measures at 6 months and 12months | baseline (early injury), post-traumatic for 6 months and 12 months
  The changes of brain volume (mm3) are evaluated by structural MRI
Change from baseline brain function measures at 6 months and 12months | baseline (early injury), post-traumatic for 6 months and 12 months
  The changes of brain functional connectivity intensity are evaluated by functional MRI

SECONDARY OUTCOMES:
Changes from baseline cognitive condition at 6 months and 12months | baseline (early injury), post-traumatic for 6 months and 12 months
  The cognitive condition is assessed by Wechsler Intelligence Scale for Children-IV-Chinese Version (WISC-IV), higher scores represent better cognitive.
Changes from baseline behavior condition at 6 months and 12months | baseline (early injury), post-traumatic for 6 months and 12 months
  the neuro-behavior condition is assessed by child behavior checklist（CBCL），higher scores represent better behavior symptoms.
Changes from baseline gut microbiota at 6 months and 12months | baseline (early injury), post-traumatic for 6 months and 12 months
  Fecal samples were collected within 2 days before or after MR examination

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China